CLINICAL TRIAL: NCT01590173
Title: Addition of Prednisolone and Heparin in Patients With Repeated Implantation Failures: a Prospective Clinical Study
Brief Title: Addition of Prednisolone and Heparin in Patients Undergoing IVF With Failed IVF Cycles
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Siristatidis Charalampos, MD, PhD, Senior Lecturer, Director of the IVF Unit, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123123
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Infertility
Keywords: Low molecular weight heparin; Prednisolone; Glucocorticoids; Recurrent implantation failure; Pregnancy rate
MeSH Terms: conditions — Infertility | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Prednisolone and Heparin during COH for IVF (Experimental)
  Interventions: Drug: Prednisolone and Heparin during COH for IVF
- COH for IVF (Active Comparator)
  Interventions: Drug: COH for IVF

INTERVENTIONS:
Drug: Prednisolone and Heparin during COH for IVF — Low Molecular Weight Heparin (LMWH) (Enoxaparin Sodium, Clexane, Sanofi-Aventis, Australia) at a dose of 1 mg/kg/day and 5 mg prednisolone p.os (Prezolon; Nycomed Hellas SA) were to be initiated on the first day of injections in both protocols until the pregnancy test. In cases of pregnancy, prednisolone and enoxaparin were to be continued up to the 12th and 34th week, respectively
  Arms: Prednisolone and Heparin during COH for IVF
Drug: COH for IVF — Both GnRH agonists (long, starting at day 2 or 21) with Triptorelin acetate 0.1 mg (Gonapetpyl daily; Ferring, Kiel, Germany) and antagonists' with ganirelix 0.25 mg (Orgalutran; Organon, Oss, The Netherlands) or cetrorelix 0.25 mg (Cetrotide; Serono, Rome, Italy) protocols will be used; for ovarian stimulation both recombinant FSH (Puregon; Organon, Oss, Netherlands or Gonal F; Serono, Rome, Italy) and human menopausal gonadotrophin (Menopur; Ferring Pharmaceuticals, Langley, Berkshire, UK) will be used. Ovarian response will be monitored by ultrasonography, oocyte retrieval will be performed 36-38 hours after the hCG triggering and for luteal phase support 600 mg progesterone tablets (Utrogestan; Laboratoires Besins- Iscovesco, Paris, France) or gel 8% intravaginally (Vasclor; Verisfield Ltd, UK) will be applied.
  Arms: COH for IVF

SUMMARY:
The addition of heparin and prednisolone increases pregnancy outcome parameters in women undergoing In Vitro Fertilisation (IVF) with failed IVF cycles.

ELIGIBILITY:
Inclusion Criteria:

* personal history of ≥2 failed IVF/ICSI cycles
* age <45 years
* availability of fresh ejaculate sperm for IVF/ICSI procedures
* confirmation of normal uterine cavity
* presence of good quality (Grade I or II) embryos for transfer

Exclusion Criteria:

* endocrine disorders
* immune disorders
* coagulation disorders

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2012-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | finding of a fetal heart at >6 gestational weeks / 2 years

SECONDARY OUTCOMES:
miscarriage rate | through study completion, an average of 2 years
live birth rate | through study completion, an average of 2 years
biochemical pregnancy rate | through study completion, an average of 2 years
OHSS | through study completion, an average of 2 years
multiple pregnancy rate | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Siristatidis, MD, PhD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Assisted Reproduction Unit, 3rd Department of Obstetrics & Gynecology, Athens, Chaidari, Attica, Greece

REFERENCES:
- [Background] Urman B, Ata B, Yakin K, Alatas C, Aksoy S, Mercan R, Balaban B. Luteal phase empirical low molecular weight heparin administration in patients with failed ICSI embryo transfer cycles: a randomized open-labeled pilot trial. Hum Reprod. 2009 Jul;24(7):1640-7. doi: 10.1093/humrep/dep086. Epub 2009 Apr 8. PMID 19357135
- [Background] Boomsma CM, Keay SD, Macklon NS. Peri-implantation glucocorticoid administration for assisted reproductive technology cycles. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD005996. doi: 10.1002/14651858.CD005996.pub2. PMID 17253574
- [Background] Nelson SM, Greer IA. The potential role of heparin in assisted conception. Hum Reprod Update. 2008 Nov-Dec;14(6):623-45. doi: 10.1093/humupd/dmn031. Epub 2008 Aug 12. PMID 18701511
- [Background] Primi MP, Senn A, Montag M, Van der Ven H, Mandelbaum J, Veiga A, Barri P, Germond M. A European multicentre prospective randomized study to assess the use of assisted hatching with a diode laser and the benefit of an immunosuppressive/antibiotic treatment in different patient populations. Hum Reprod. 2004 Oct;19(10):2325-33. doi: 10.1093/humrep/deh430. Epub 2004 Jul 29. PMID 15284215